CLINICAL TRIAL: NCT06081218
Title: Effect of Acute Exercise on Cognitive Functions and Blood Markers of Brain Plasticity in Regular Chronic Cannabis Users
Acronym: CANNABEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016_70
Record Dates: First submitted 2023-07-06; First posted 2023-10-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Cannabis User
MeSH Terms: interventions — Carcinogenicity Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic cannabis users (Experimental)
  Interventions: Other: activity test
- Healthy subjects (Sham Comparator)
  Interventions: Other: activity test

INTERVENTIONS:
Other: activity test — Over 2 weeks, participants have to do a maximal progressive exercise and a 30 min constant exercise at 50% of maximal aerobic power

SUMMARY:
The endocannabinoid system (ECS) is a complex endogenous signaling system made up of transmembrane cannabinoid receptors (CB1 and CB2 receptors), their endogenous lipid-derived ligands (the endocannabinoids - eCBs), and enzymes for ligand biosynthesis and degradation. Interestingly, exercise increase plasma AEA, one of the most famous endocannabinoid. This increase could be involved in exercise-induced neurogenesis and other beneficial exercise adaptations. Chronic cannabis use is associated with alteration of ECS activity. The aim of the study is to compare ECS response to exercise between chronic cannabis users and non-users.

ELIGIBILITY:
Inclusion Criteria:

Cannabis consumer group:

* Cannabis consumption > 100 times in lifetime, last exposure < 7 days, and recent exposure > 10 times in the month.
* Positive toxicological urine test for ∆-9-THC.
* Having a cannabis use disorder according to the CAST.

Healthy group:

* Negative urine toxicological test for cannabis.
* No regular cannabis use for more than 6 months once in a lifetime.
* No cannabis consumption in the 6 months preceding the study.

Exclusion Criteria:

For all subjects :

* Disorders of use of other substances (alcohol, cocaine, opioid, or synthetic drugs).
* Alcohol consumption greater than 30g per day (averaged over one week) and/or alcohol abuse the week preceding the visit.
* Under medical treatment.
* Presence of diagnosed neurological disorders.
* Diagnosis of a psychotic picture entering axis I, DSM-5.
* Chronic progressive disease or in remission.
* Body mass index > 30 kg/m2 (i.e. presence of obesity).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma endocannabinoids levels (pmol/ml) | 2 weeks

SECONDARY OUTCOMES:
regulating hormone of endocannabinoids (plasma levels of cortisol, ng/ml) | 2 weeks
Blood marker of neurogenesis and neuroplasticity (plasma levels and BDNF, pg/ml) | 2 weeks
change in cerebral muscular, oxygenation (HHB), (HbO2), (Hbtot) (arbitrary unit) | 2 weeks
Cognitive function (selective attention, stroop test) | 2 weeks
  The stroop test can be used to measure a person's selective attention capacity
Oxygen consumption (VO2) (ml/min/kg) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Lille, Lille, France